CLINICAL TRIAL: NCT01930214
Title: Multi-center Prospective Study to Evaluate Outcomes of the Moderate to Severely Calcified Coronary Lesions (MACE)
Acronym: MACE
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-0002-P
Record Dates: First submitted 2013-08-21; First posted 2013-08-28 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- None/mild calcification: Presence of readily apparent radiopacities within the vascular wall at the site of the stenosis.
  Interventions: Device: Percutaneous Coronary Intervention
- Moderate Calcification: Presence of radiopacities only during the cardiac cycle before contrast injection with calcium extended partially into the target lesion.
  Interventions: Device: Percutaneous Coronary Intervention
- Severe calcification: Presence of radiopacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location, total length of calcium (including segmented) must be at least 15mm and extend partially into the target lesion.
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Any Food and Drug Administration (FDA) commercially available device for treating none/mild, moderate, and severe calcified coronary lesions, with the exception of CSI's Coronary Orbital Atherectomy System (OAS).

SUMMARY:
The objective of this study is to assess the current standard of care treatment outcome in none/mild, moderate and severely calcified coronary lesions using:

* A composite of MACE at 30-day and one (1) year post procedure, and
* Procedural and lesion success

DETAILED DESCRIPTION:
This prospective, non-randomized, multi-center study includes subjects who meet all of the inclusion and none of the exclusion criteria and sign the ICF. This study may treat up to approximately 500 subjects at up to 50 active sites in the U.S. Subjects may be followed up to three (3) years. Subjects will be stratified into one (1) of three (3) arms based on the degree of calcification in the coronary lesion as defined by this protocol. The duration of the study is expected to be approximately four (4) years.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age.
2. Subjects must be scheduled for percutaneous coronary revascularization involving stent deployment in de novo coronary lesions. Percutaneous coronary revascularization is defined as treatment with commercially available devices that may include but not limited to balloon angioplasty, cutting balloon, rotablation, etc. followed by the stent placement.
3. Subjects CK-MB must be less than or equal to the upper limit of lab normal value within eight (8) hours prior to procedure. If CK-MB results are not yet available prior to initiating procedure, subjects Troponin I or Troponin T must be less than or equal to the upper limit of lab normal value within eight (8) hours prior to the procedure.
4. The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure.
5. The target vessel must be a native coronary artery with:

   1. A stenosis ≥ 70% and < 100%, or
   2. A stenosis ≥ 50% < 70% with evidence of clinical ischemia
6. The target vessel reference diameter must be ≥ 2.5mm and ≤ 4.0 mm.
7. The lesion length must not exceed 40 mm.
8. The target vessel must have a Thrombolysis In Myocardial Infarction (TIMI) flow three (3) at baseline.

Exclusion Criteria:

1. Inability to understand the study or a history of non-compliance with medical advice.
2. Unwilling or unable to sign the MACE clinical study ICF.
3. History of any cognitive or mental health status that would interfere with study participation.
4. Currently enrolled in any other pre-approval investigational study. This does not apply to long-term post-market studies unless these studies might clinically interfere with the current study endpoints (e.g., limit use of study-required medication, etc.).
5. Female subjects who are pregnant or planning to become pregnant within the study period.
6. Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine or clopidogrel without adequate alternative medications.
7. Known sensitivity to contrast media, which cannot be adequately pre-medicated.
8. Diagnosed with chronic renal failure unless under hemodialysis, or has a serum creatinine level >2.5 mg/dl.
9. History of major cardiac intervention within 30-day, not including a PCI procedure for a staging purpose.
10. Evidence of heart failure by one of the following:

    i. Left Ventricular Ejection Fraction (LVEF) ≤ 25% ii. New York Heart Association (NYHA) class III or IV iii. Clinical symptoms
11. History of a stroke or transient ischemic attack (TIA) within six (6) months
12. Active peptic ulcer or upper gastrointestinal (GI) bleeding within six (6) months.
13. History of bleeding diathesis or coagulopathy or intention to refuse blood transfusion if one should become necessary.
14. Concurrent medical condition with a life expectancy of < 36 months.
15. History of immune deficiency.
16. Uncontrolled insulin dependent diabetes.
17. Evidence of active infections on the day of the index procedure.
18. Subject has planned cardiovascular intervention within 60 days post index procedure.
19. Subject with angiographically confirmed evidence of more than two (2) lesions within one (1) vessel or more than one (1) vessel requiring intervention, unless the treatment is staged. See Section 10.1 for more details.
20. Target lesion is located in a native vessel distal to anastomosis with a saphenous vein graft or Left Internal Mammary Artery/ Right Internal Mammary Artery (LIMA/RIMA) bypass.
21. Target vessel has angiographically visible or suspected thrombus.
22. Target vessel appears to be/is excessively tortuous at baseline.
23. Target lesion is an ostial location (within 5mm of ostium) or an unprotected left main lesion.
24. Target lesion is a bifurcation (side branch ≥ 1.5mm).
25. Treatment of the target lesion with the CSI coronary Diamondback Orbital Atherectomy System (OAS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years or older who are scheduled for percutaneous coronary revascularization involving stent.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samin K Sharma, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (34):
- United States (34):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Glendale Adventist Medical Center, Glendale, California
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital, Washington D.C., District of Columbia
  - Clearwater Cardiovascular & Interventional Consultants, Clearwater, Florida
  - Mount Sinai Medical Center Heart Institute, Miami Beach, Florida
  - Cardiovascular Institute of NW Florida, Panama City, Florida
  - Georgia Regents Research Institute, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - John Hopkins, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - McLaren Bay Regional, Bay City, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Boone Hospital, Columbia, Missouri
  - Saint Luke's, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Mount Sinai New York, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - North Carolina Heart & Vascular Specialists, Raleigh, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - St. John Health System, Tulsa, Oklahoma
  - University Pittsburg MC - Hamot, Erie, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
  - Mission Research Institute, New Braunfels, Texas
  - Providence Health Center, Waco, Texas

REFERENCES:
- [Result] Sharma SK, Bolduan RW, Patel MR, Martinsen BJ, Azemi T, Giugliano G, Resar JR, Mehran R, Cohen DJ, Popma JJ, Waksman R. Impact of calcification on percutaneous coronary intervention: MACE-Trial 1-year results. Catheter Cardiovasc Interv. 2019 Aug 1;94(2):187-194. doi: 10.1002/ccd.28099. Epub 2019 Jan 25. PMID 30681262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was completed at 350 treated subjects.
Pre-assignment Details: A subject was considered enrolled when a signed informed consent was in place, all inclusion/no exclusion criteria were met, and the study guidewire had crossed the target lesion.
Period: Overall Study
Arm/Group | None/Mild Calcification | Moderate Calcification | Severe Calcification
Started | 100 | 117 | 133
Completed | 80 | 96 | 108
Not Completed | 20 | 21 | 25
Not completed — Death | 4 | 4 | 11
Not completed — Lost to Follow-up | 12 | 13 | 12
Not completed — Voluntary withdrawal of infomed consent | 2 | 4 | 2
Not completed — Physician Decision | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population summarizes data from 350 enrolled subjects. Outcome Measures data includes the 346 subjects with sufficient angiography for core lab stratification.
Groups:
- Total: Total of all reporting groups
Arm/Group | None/Mild Calcification | Moderate Calcification | Severe Calcification | Total
Number analyzed (Participants) | 100 | 117 | 133 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.3) | 68.9 (10.6) | 69.3 (9.2) | 67.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 34 | 92
  Male | 71 | 88 | 99 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 5 | 19
  Not Hispanic or Latino | 94 | 109 | 128 | 331
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 88 | 98 | 118 | 304
  Black or African American | 9 | 13 | 6 | 28
  Asian | 3 | 5 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Native American | 0 | 1 | 0 | 1
  Other | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 100 | 117 | 133 | 350

OUTCOME MEASURES:

1. Primary Outcome: MACE at 30 Days
Description: A Kaplan-Meier analysis was performed to determine the percent probability that a study participant experienced a major adverse cardiac event through 30 days.
  30-day MACE is composed of:
  * Cardiac death
  * Myocardial Infarction (MI) - defined as a Creatine Kinase Myocardial-Band Isoenzyme (CK-MB) level greater than three (3) times the Upper Limit of Lab Normal (ULN) value with or without new pathologic Q wave
  * Target Vessel Revascularization (TVR) - defined as a revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure
Time Frame: 30 days post procedure
Population: Subjects were enrolled based on Investigator assessment of calcium; however, all analyses were performed by core lab assessed calcium to ensure consistent methodology. Of the 350 subjects enrolled in the study, 346 had sufficient angiography for core lab stratification (133 none/mild, 99 moderate, and 114 severe).
Measure: Number (95% Confidence Interval); unit: Percent probability of MACE
Groups:
- None/Mild Calcification: Presence of readily apparent radiopacities within the vascular wall at the site of the stenosis as assessed by the angiographic core lab.
  Percutaneous Coronary Intervention: Any Food and Drug Administration (FDA) commercially available device for treating none/mild, moderate, and severe calcified coronary lesions, with the exception of CSI's Coronary Orbital Atherectomy System (OAS).
- Moderate Calcification: Presence of radiopacities only during the cardiac cycle before contrast injection with calcium extended partially into the target lesion as assessed by the angiographic core lab.
  Percutaneous Coronary Intervention: Any Food and Drug Administration (FDA) commercially available device for treating none/mild, moderate, and severe calcified coronary lesions, with the exception of CSI's Coronary Orbital Atherectomy System (OAS).
- Severe Calcification: Presence of radiopacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location, total length of calcium (including segmented) must be at least 15mm and extend partially into the target lesion as assessed by the angiographic core lab.
  Percutaneous Coronary Intervention: Any Food and Drug Administration (FDA) commercially available device for treating none/mild, moderate, and severe calcified coronary lesions, with the exception of CSI's Coronary Orbital Atherectomy System (OAS).
Arm/Group | None/Mild Calcification | Moderate Calcification | Severe Calcification
Number analyzed (Participants) | 133 | 99 | 114
Percent probability of MACE | 2.3 [0.0 to 4.8] | 3.1 [0.0 to 6.5] | 15 [8.4 to 21.6]

2. Secondary Outcome: MACE at One (1) Year
Description: A Kaplan-Meier analysis was performed to determine the percent probability that a study participant experienced a major adverse cardiac event through 1 year.
  1-year MACE is composed of:
  * Cardiac death
  * Myocardial Infarction (MI) - defined as a Creatine Kinase Myocardial-Band Isoenzyme (CK-MB) level greater than three (3) times the Upper Limit of Lab Normal (ULN) value with or without new pathologic Q wave
  * Target Vessel Revascularization (TVR) - defined as a revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure
Time Frame: One (1) year post procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent probability of MACE
Arm/Group | None/Mild Calcification | Moderate Calcification | Severe Calcification
Number analyzed (Participants) | 133 | 99 | 114
Percent probability of MACE | 5.4 [1.5 to 9.2] | 8.5 [2.8 to 14.2] | 24.2 [16.1 to 32.4]

3. Secondary Outcome: Procedural Success
Description: Procedural success is defined as success in facilitating stent delivery with a residual stenosis of <50% and without the occurrence of an in-hospital MACE.
Time Frame: Participants were followed from baseline procedure through hospital discharge, an expected average of 24 hours
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent of Procedures
Arm/Group | None/Mild Calcification | Moderate Calcification | Severe Calcification
Number analyzed (Participants) | 133 | 99 | 114
Percent of Procedures | 97.7 [93.5 to 99.5] | 96 [90.0 to 98.9] | 86.8 [79.2 to 92.4]

4. Secondary Outcome: Lesion Success
Description: Lesion success is defined as success in facilitating stent delivery with a post-procedural result of <50% residual stenosis for a given lesion treated during the procedure without severe angiographic complications.
Time Frame: During the procedure
Population: as for outcome 1
Measure: Number; unit: Percentage of Procedures
Arm/Group | None/Mild Calcification | Moderate Calcification | Severe Calcification
Number analyzed (Participants) | 133 | 99 | 114
Percentage of Procedures | 94.7 | 88.9 | 83.3

ADVERSE EVENTS:
Time Frame: 3 years
Description: AE collection was limited to cardiac event, death, serious injury, MAEs, bleeding and angio complications related to the index procedure. Angio core lab (CL) assessed the presence of dissections and perforations; CEC adjudicated: bleed, angio events not assessed by CL, death, MI, TVR, TLR and any non-endpoint event that the CEC deemed necessary to adjudicate as study related. Groups based on CL calcification for 346/350; remaining (4) subjects were included based on site reported calcification.
Groups:
- None/Mild Calcification: • Presence of readily apparent radiopacities within the vascular wall at the site of the stenosis.
  Percutaneous Coronary Intervention: Any Food and Drug Administration (FDA) commercially available device for treating none/mild, moderate, and severe calcified coronary lesions, with the exception of CSI's Coronary Orbital Atherectomy System (OAS).
- Moderate Calcification: • Presence of radiopacities only during the cardiac cycle before contrast injection with calcium extended partially into the target lesion.
  Percutaneous Coronary Intervention: Any Food and Drug Administration (FDA) commercially available device for treating none/mild, moderate, and severe calcified coronary lesions, with the exception of CSI's Coronary Orbital Atherectomy System (OAS).
- Severe Calcification: • Presence of radiopacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location, total length of calcium (including segmented) must be at least 15mm and extend partially into the target lesion.
  Percutaneous Coronary Intervention: Any Food and Drug Administration (FDA) commercially available device for treating none/mild, moderate, and severe calcified coronary lesions, with the exception of CSI's Coronary Orbital Atherectomy System (OAS).
Arm/Group | None/Mild Calcification | Moderate Calcification | Severe Calcification
All-Cause Mortality (participants affected / at risk) | 6/134 | 1/99 | 7/117
Serious Adverse Events (participants affected / at risk) | 62/134 | 47/99 | 64/117
Other Adverse Events (participants affected / at risk) | 0/134 | 0/99 | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | None/Mild Calcification (N=134) | Moderate Calcification (N=99) | Severe Calcification (N=117)
Acute MI, Q-wave (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute MI, non Q-wave (Cardiac disorders) | 9 (9) | 6 (7) | 17 (19)
Acute congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 17 (23) | 10 (14) | 12 (21)
Arrhythmia, unspecified (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 5 (5) | 4 (5) | 5 (5)
Atrioventricular block, III degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 8 (8) | 3 (3) | 1 (1)
Chest Pain, non ischemic (Cardiac disorders) | 6 (6) | 3 (3) | 4 (4)
Chronic CHF, or exacerbation (Cardiac disorders) | 3 (4) | 3 (4) | 3 (3)
Coronary artery restenosis (Cardiac disorders) | 2 (3) | 1 (1) | 9 (13)
Elevated CK-MB (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Elevated Troponin (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Elevated cardiac enzymes (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Other cardiovascular system related AE (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abrupt or threatened closure of coronary artery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) — Angiographic complications
Coronary artery vasospasm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Angiographic complications
Coronary vessel dissection present (A-F) (Injury, poisoning and procedural complications) | 12 (12) | 16 (16) | 25 (25) — Angiographic complications
Coronary vessel perforation present (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) — Angiographic complications
Slow flow or no reflow phenomena (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) — Angiographic complications
Deep vein thrombosis (DVT) (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hematoma at access site, not requiring intervention (Vascular disorders) | 3 (3) | 3 (3) | 2 (2)
Hemorrhage, major, requiring transfusion (Vascular disorders) | 1 (1) | 0 (0) | 4 (4)
Hemorrhage, minor, without transfusion (Vascular disorders) | 4 (4) | 3 (4) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 1 (1)
Peripheral artery pseudoaneurysm (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Peripheral artery/vascular disease (Vascular disorders) | 2 (2) | 3 (4) | 0 (0)
Peripheral vessel damage requiring surgical repair (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (CVA) (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnea/Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Renal insufficiency (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Allergic reaction to contrast dye (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (General disorders) | 1 (1) | 0 (0) | 3 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infection, systemic (General disorders) | 1 (1) | 0 (0) | 1 (1)
Other index procedure related AE (General disorders) | 0 (0) | 1 (1) | 0 (0)
Other infection (General disorders) | 2 (2) | 0 (0) | 0 (0)
Other patient condition related AE (General disorders) | 3 (3) | 2 (2) | 4 (4)
Trauma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Death (General disorders) | 2 (2) | 1 (1) | 4 (4)
Cardiac Death (Cardiac disorders) | 4 (4) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any previously unpublished information provided to the Investigators by the Sponsor is confidential and will remain the sole property of the Sponsor. The Investigator agrees to use this information only in accomplishing this study not use it for other purposes without the Sponsor's written consent. An Investigator can generate additional publication ideas based on the trial data. The Sponsor reserves the right to review the manuscript prior to submission in order to verify accuracy of the data